# Study Protocol and Statistical Analysis Plan (SAP) — Frailty Evaluation Component

#### 1. Administrative information

Study title (short): FRAGSALUD — educational programme for frail/pre-frail older adults.

ClinicalTrials.gov Identifier: NCT05610605.

Study period: Conducted March 2022 – September 2023; assessments at baseline, 6 months (end of intervention), and 12 months (6 months post-intervention).

Primary SAP scope: frailty phenotype (Fried criteria) — score, categorical status (robust / pre-frail / frail).

Document date: 24/09/2025

#### 2. Background & rationale (frailty)

Frailty is a state of increased vulnerability to stressors reflecting reduced physiological reserve. The study tested whether a 6-month educational intervention changes frailty status and frailty score compared with usual care in community-dwelling older adults with at least one Fried criterion.

## 3. Objectives (frailty component)

Primary frailty objective: Evaluate the effect of the 6-month educational programme on the Fried frailty total score at 6 months (end of intervention) and at 12 months (6 months post-intervention), compared with control.

Secondary frailty objectives:

- Evaluate shifts in frailty categories (robust / pre-frail / frail) between baseline, 6 months and 12 months.

## 4. Study design (brief)

Multicentre, parallel-group randomised controlled trial; participants randomised to educational programme or control (usual care). Assessments at baseline, 6 months, and 12 months.

# 5. Population and eligibility

Inclusion: Community-dwelling adults aged  $\geq$ 65 years with  $\geq$ 1 Fried frailty criterion (prefrail or frail).

Exclusion: Institutionalised individuals; robust participants (zero Fried criteria).

Final analysed sample: 199 participants (109 intervention, 90 control after attrition).

## 6. Frailty measurement (operational definition)

Frailty was operationalised using the Fried physical frailty phenotype, consisting of:

- Shrinking (unintentional weight loss  $\geq$ 4.5 kg or  $\geq$ 5% in past year).
- Weakness (sex- and BMI-specific grip strength cut-offs).
- Poor endurance/exhaustion (self-reported ≥3 days in previous week).
- Slowness (4-m timed walk with sex- and height-specific cut-offs).
- Low physical activity (Minnesota Leisure Time Physical Activity Questionnaire).

Scoring: 0–5. Categories: robust = 0; pre-frail = 1–2; frail  $\geq$ 3.

## 7. Outcomes (frailty-specific)

Primary frailty outcome: Change in Fried total score from baseline to 6 months and 12 months.

Secondary frailty outcomes:

- Proportion of participants in each frailty category at each timepoint.

### 8. Sample size

Target  $\geq$ 196 participants, based on effect size 0.5 SD,  $\alpha$  = 0.05, power = 80%, allowing for 15% dropout.

#### 9. Randomisation and allocation

Computerised block randomisation ensuring balance between groups.

#### 10. Blinding

Participants and intervention deliverers were not blinded. Outcome assessors and analysts were blinded where possible.

#### 11. Data collection schedule

Baseline: Fried components.

6 months: repeat assessments.

12 months: repeat assessments.

# 12. Statistical Analysis Plan

Analysis populations: Intention-to-treat and per-protocol (sensitivity).

Primary analysis: Linear mixed-effects model with Fried score as dependent variable; fixed effects for group, time, and group × time; random effect for participant; adjusted for age, sex, education.

Secondary analysis: Frailty category transitions using chi-square, logistic regression, or multinomial models.

Sensitivity analyses: per-protocol, alternative frailty scoring, responder definitions.

# 13. Reporting and tables/figures

Baseline frailty table by arm.

Adjusted change table with  $\beta$  (95% CI) and p-values.

Frailty category transitions figure.

# 14. Key frailty results

At 6 months, intervention group reduced Fried score by -0.60 vs -0.015 in controls ( $\beta = -0.515$ , p = 0.007).

At 12 months,  $\beta = -0.714$ , p < 0.001.

Frailty category improved in intervention group: increase in robust participants, reduction in frail participants.